CLINICAL TRIAL: NCT01275482
Title: Effectiveness of Transverse Friction Massage Causing or Not Local Twitch Response in Anterior Deltoid Muscle Latent Myofascial Trigger Points
Brief Title: Effectiveness of Transverse Friction Massage in Latent Myofascial Trigger Points in Anterior Deltoid Muscle
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Jose Miota, University of Castilla-La Mancha
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: deltoid
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Myofascial Trigger Points; Myofascial Pain
Keywords: Latent Myofascial trigger point.; Transverse friction massage; Local twitch response; Effectiveness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- isolated contractions caused (Experimental): The investigators do TFM causing isolated contractions in de muscle fibers containing de latent trigger point.
  Interventions: Procedure: Transverse friction massage (TFM)
- No isolated contraction caused (Active Comparator): The investigators don´t cause contraction during the TFM
  Interventions: Procedure: Transverse friction massage (TFM)

INTERVENTIONS:
Procedure: Transverse friction massage (TFM) — The TFM was describe of Cyriax as an effective method to treat soft tissues. It is a massage done always in perpendicular direction of damage tissue. During the massage, we can caused isolated contractions from the fiber muscles containing the latent trigger points.
  Other Names: Cyriax massage
  Arms: isolated contractions caused
Procedure: Transverse friction massage (TFM) — The TFM was describe of Cyriax as an effective method to treat soft tissues. It is a massage done always in perpendicular direction of damage tissue.
  Other Names: Cyriax massage

SUMMARY:
The purpose of this study is to determine whether Transverse Friction Massage (TFM) in Latent Myofascial Trigger points (MTrP) is more effective making this technique in two different ways.

DETAILED DESCRIPTION:
The investigators divide in two groups. The investigators apply the TFM in similar way in both, but the investigators cause local twitch response (isolated contraction of muscle fibers containing the latent trigger points)just in one group. So the investigators want to know whether the effectiveness of this technique is due to those local twitch responses, comparing both groups. The investigators asses Strength, range of motion, and overall, pressure pain thresholds to evaluate the pain sensitivity progress.

ELIGIBILITY:
Inclusion Criteria:

* Having latent myofascial trigger points in anterior deltoid
* Visual local twitch response

Exclusion Criteria:

* Having active Myofascial trigger points in anterior deltoid
* Having suffered injuries or surgery in upper limb.
* Pain in the first evaluation session.
* Not obtaining local twitch response

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pressure pain Threshold (PPT)during treatment. | Pre and post treatment every session and 1 week after last session
  The PPT is defined as the minimal amount of pressure where a sense of pressure first changes to discomfort or pain in a certain point

CONTACTS AND LOCATIONS:
Overall Officials: Jose Miota, PhT, Principal Investigator — UCastilla-La Mancha
Locations (1):
- UCLM, Toledo, Toledo, Spain